CLINICAL TRIAL: NCT04402229
Title: Psychological Impact of the Covid-19 Pandemic on Student Nurses :Prevalence and Risk Factors of Acute Post-traumatic Stress Symptoms 1 Month After the Epidemic Peak
Brief Title: Psychological Impact of the Covid-19 Pandemic on Student Nurses
Acronym: StudentCov
Status: Completed | Type: Observational
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Jacq Gwenaelle, Investigator Coodinator, Versailles Hospital
Other Study IDs: P17/04_StudentCov
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Nurse; Student; Post Traumatic Stress Disorder; COVID-19
Keywords: student nurses; covid-19; post tramatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The World Health Organization (WHO) declared in early 2020 the emergence of a new highly contagious SARS-CoV-2 coronavirus responsible for a global public health emergency. In France, the first cases of contamination have been reported since the end of January 2020, and the first death in mid-February 2020. Then, data published by Public Healh France reported an increasing and rapidly exponential number of contaminations. First cases have been identified on a cluster mode, then rapidly spreading in some French departments and regions, indicating rapid kinetics of virus spread. Given the magnitude of the situation both French territory and neighboring European territories (mainly Italy), the government mobilized the entire health system to critically manage this epidemic. This exceptional and unprecedented pandemic deeply impacted the health structures, disrupting healthcare organizations. All caregivers, including all student nurses, actively participated in the mobilization and strengthening of care teams. The health crisis exposed the population of caregivers to potentially traumatic events which can have major repercussions on their health state. The description and identification of the risk factors of the occurrence of post traumatic stress disorders in student nurses during the health crisis would allow to provide avenues for improving training devices and to facilitate health workers access to specific psychological care particularly dedicated to the student nurses population needs.

DETAILED DESCRIPTION:
Describe the prevalence of post-traumatic stress disorder among student nurses 1 month after the end of the French epidemic Covid-19 peak

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old

Exclusion Criteria:

* Opposition to participate to the questionnaire

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All French Student Nurses
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of PTSD-related symptoms assessed by the IES-R | 1 month after the end of the French epidemic Covid-19 peak
  Proportion of students with IES-R> 22 PTSD-related symptoms. Impact of Event Scale - Revised (IES-R) is a 22-item self-report measure that assesses subjective distress caused by traumatic events. ... The IES-R yields a total score (ranging from 0 to 88) and subscale scores can also be calculated for the Intrusion, Avoidance, and Hyperarousal subscales.

SECONDARY OUTCOMES:
PTSD-related symptoms assessed by the IES-R in the total population of students nurses | 1 month after the end of the French epidemic Covid-19 peak
  IES-R> 22 PTSD-related symptoms in the total population of students nurses( 3 years training)
PTSD-related symptoms assessed by the IES-R according to student's years of school | 1 month after the end of the French epidemic Covid-19 peak
  IES-R> 22 PTSD-related symptoms in each population of students nurses of first-, second-, and third-year.

CONTACTS AND LOCATIONS:
Overall Officials: Gwenaelle Jacq, RN, Principal Investigator — CH Versailles
Locations (2):
- France (2):
  - Versailles hospital, Le Chesnay
  - Toulouse University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No